CLINICAL TRIAL: NCT03003676
Title: A Pilot Study of Sequential ONCOS-102, an Engineered Oncolytic Adenovirus Expressing GMCSF, and Pembrolizumab in Patients With Advanced or Unresectable Melanoma Progressing After PD1 Blockade
Brief Title: A Pilot Study of Sequential ONCOS-102, an Engineered Oncolytic Adenovirus Expressing GMCSF, and Pembrolizumab in Patients With Advanced or Unresectable Melanoma Progressing After Programmed Cell Death Protein 1 (PD1) Blockade
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Targovax Oy (Industry)
Responsible Party: Sponsor
Organization: Targovax ASA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONCOS C824
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-07

CONDITIONS: Advanced or Unresectable Melanoma Progressing After PD1 Blockade
MeSH Terms: interventions — Cyclophosphamide; pembrolizumab

ARMS (1):
- Experimental: ONCOS-102+cyclophosphamide+pembrolizumab (Experimental): Part I: Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will then receive pembrolizumab i.v., 2mg/kg or 200mg flat dose, on day 22 (Week 3) and every 3 weeks thereafter until the end of treatment visit on day 169 (Week 24).
  Part II: Patients will receive 4 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, 8 and 15) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. ONCOS-102 will be given in combination with Pembrolizumab starting on Day 22/Week 3 and every three weeks thereafter until Day 169/Week 24 or until unacceptable toxicity or clinically relevant disease progression, whichever occurs first. Pembrolizumab will be given according to institutional practice (2mg/kg or 200mg flat dose).
  Interventions: Biological: ONCOS-102; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Biological: ONCOS-102 — Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
Drug: Cyclophosphamide — Pre-treatment
Drug: Pembrolizumab — PD1 blockade

SUMMARY:
This is a multi center, phase I pilot study of sequential ONCOS-102 and pembrolizumab in patients with advanced or unresectable melanoma progressing after PD1 blockade. The primary objective of the study is to determine the safety of sequential treatment with ONCOS-102 followed by pembrolizumab. The protocol aims to enroll patients into two cohorts: Part I: up to 12 patients will receive sequential treatment with ONCOS-102 followed by pembrolizumab. Part II: up to 12 patients will receive an initial treatment phase with ONCOS-102 followed by a treatment phase with ONCOS-102 in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* For US sites: Histopathologically confirmed melanoma with an injectable cutaneous or lymph node metastasis that has progressed in the opinion of the treating investigator despite administering a Food and Drug Administration (FDA) approved anti-PD1 agent, with or without ipilimumab.
* For European sites: Histopathologically confirmed melanoma with an injectable cutaneous or lymph node metastasis that has progressed in the opinion of the treating investigator despite administering a regulatory approved anti-PD1 agent, with or without ipilimumab.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
* Measurable disease according to RECIST 1.1.
* Acceptable coagulation status: international normalised ratio (INR) of blood clotting, prothrombin time and activated partial thromboplastin time within ≤1.5 x upper limit of normal (ULN).
* Completion of local therapy, such as radiation, surgical resection, injectable immunebased therapy, or topical pro-inflammatory agent, 21 days prior to first dose of protocol therapy.
* Adverse events from previous cancer therapies (excluding alopecia) must have recovered to grade 1 (CTCAE, most recent version). Stable grade 2 AEs such as endocrine conditions are allowed, and other chronic stable AEs may be considered on a case by case basis by the Principal Investigator.
* Clinical stability of brain metastases for at least 4 weeks prior to first day of study therapy.
* Acceptable liver and renal functions defined as:

  * Total bilirubin ≤1.5 x ULN (does not include patients with Gilbert's Disease)
  * Aspartate aminotransferase (AST, SGOT), alanine aminotransferase (ALT, SGPT) ≤3.0 x ULN
  * Serum creatinine ≤1.5 x ULN
* Acceptable haematological function defined as (Patients can be transfused to meet the haemoglobin entry criteria):

  * Haemoglobin ≥9 g/dL
  * Neutrophils ≥1.5 x 10^9/L
  * Platelet count ≥75 x 10^9/L
* Able to provide valid written informed consent.
* All women of childbearing potential must have a negative urine or serum pregnancy test at screening.
* For US sites: All patients must agree to use barrier contraception (i.e. condom) during study treatment and for 2 months after the last virus treatment and 4 months after the last dose of chemotherapy and pembrolizumab.
* For European sites: All patients must agree to use highly effective contraception for at least 6 months (according to the latest country specific SmPC) after administration of CPO, up to 4 months after last dose of pembrolizumab, and up to 2 months after last dose of ONCOS-102, whichever comes last.
* For European sites: All women of child-bearing potential must agree to perform pregnancy testing throughout the study starting at baseline, every 3 weeks from day 22 until last dose of study medication (ONCOS-102 and pembrolizumab) and then every month for at least 6 months.

Exclusion Criteria:

* A concomitant medical condition requiring receipt of a therapeutic anticoagulant that in the opinion of the treating physician cannot safely allow for therapeutic injection of ONCOS-102 and tumor biopsies. Local clinical practice can be followed with regard to holding a therapeutic anticoagulant during invasive procedures such as biopsies.
* A concomitant medical condition that in the opinion of the treating physician would pose unreasonable additional risk to therapeutic injection of ONCOS-102.
* For US sites: Receipt of Investigational agents within 28 days prior to first dose of protocol therapy.
* For European sites: Current participation or participation in a study of an investigational agent within 28 days prior to first dose of protocol therapy. Note: participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Any symptomatic autoimmune disease (such as lupus, scleroderma, Crohn's disease, ulcerative colitis) that requires administration of >10mg of prednisone equivalent. Lower dose steroids for conditions such as hypophysitis are allowed.
* Any prior severe adverse event attributed to prior anti-PD1 therapy that, in the Principal investigator's opinion, would contraindicate pembrolizumab administration such as:

  * Grade 2 or higher pneumonitis
  * Grade 4 AST or ALT elevation
  * Grade 3 or higher colitis attributable to PD1 blockade; note that colitis attributable to ipilimumab is not excluded
  * Note: in the absence of clinical symptoms of pancreatitis, elevations of amylase or lipase are not contraindications to therapy on this trial
* Known active infection with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or HIV. Cleared HBV/HCV infection is not an exclusion, nor is HIV infection with cluster of differentiations 4 (CD4) counts >500 and an undetectable viral load.
* Active bacterial, viral, or fungal infections, requiring systemic therapy apart from anti-viral maintenance therapy for HIV.
* History of organ transplant.
* Patients requiring chronic systemic immunosuppressants, including steroids (prednisone daily equivalent of >10 mg).
* Brain metastases that are clinically unstable (e.g. showing unequivocal growth on imaging, requiring radiation therapy, or steroids >10mg of prednisone equivalent) within 4 weeks of first dose of study drug.
* Known severe congenital or acquired cellular or humoral immunodeficiency such as common variable immunodeficiency.
* For US sites: Women who are pregnant or breast-feeding currently or are planning to conceive during or up to 4 months after end of protocol therapy.
* For European sites: Women who are currently pregnant or breast-feeding or are planning to conceive during or up to 6 months after end of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12; Primary Completion 2020-07 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - University of Maryland Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Oslo University Hospital - The Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kuryk L, Moller AW, Jaderberg M. Combination of immunogenic oncolytic adenovirus ONCOS-102 with anti-PD-1 pembrolizumab exhibits synergistic antitumor effect in humanized A2058 melanoma huNOG mouse model. Oncoimmunology. 2018 Oct 29;8(2):e1532763. doi: 10.1080/2162402X.2018.1532763. eCollection 2019. PMID 30713786

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab - Part 1: Part I: Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will receive pembrolizumab i.v., 2mg/kg or 200 mg flat dose on day 22 (Week 3) and every three weeks thereafter until Day 169/Week 24.
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab - Part 2: Part II: Patients will receive 4 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, 8 and 15) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. ONCOS-102 will be given in combination with Pembrolizumab starting on Day 22/Week 3 and every three weeks thereafter until Day 169/Week 24 or until unacceptable toxicity or clinically relevant disease progression, whichever occurs first. Pembrolizumab will be given according to institutional practice (2mg/kg or 200mg flat dose).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF) Cyclophosphamide: Pre-treatment Pembrolizumab: PD1 blockade
Period: Overall Study
Arm/Group | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab - Part 1 | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab - Part 2
Started | 9 | 12
Completed | 3 | 4
Not Completed | 6 | 8
Not completed — Lack of Efficacy | 5 | 7
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Hepatitis B infection | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1: Part I: Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will then receive pembrolizumab i.v., 2mg/kg or 200mg flat dose, on day 22 (Week 3) and every 3 weeks thereafter until the end of treatment visit on day 169 (Week 24).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2: Part II: Patients will receive 4 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, 8 and 15) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. ONCOS-102 will be given in combination with Pembrolizumab starting on Day 22/Week 3 and every three weeks thereafter until Day 169/Week 24 or until unacceptable toxicity or clinically relevant disease progression, whichever occurs first. Pembrolizumab will be given according to institutional practice (2mg/kg or 200mg flat dose).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
- Total: Total of all reporting groups
Arm/Group | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1 | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2 | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 8
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (13.68) | 67.3 (13.50) | 68.1 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18
  Norway | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events Including Treatment-emergent Serious Adverse Events Assessed by Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1: Part I1 Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will then receive pembrolizumab i.v., 2mg/kg or 200mg flat dose, on day 22 (Week 3) and every 3 weeks thereafter until the end of treatment visit on day 169 (Week 24).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2: Part 2: Patients will receive 4 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, 8 and 15) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. ONCOS-102 will be given in combination with Pembrolizumab starting on Day 22/Week 3 and every three weeks thereafter until Day 169/Week 24 or until unacceptable toxicity or clinically relevant disease progression, whichever occurs first. Pembrolizumab will be given according to institutional practice (2mg/kg or 200mg flat dose).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
Arm/Group | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1 | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2
Number analyzed (Participants) | 9 | 12
participants
  Number of patients with Treatment Emergent Adverse Event (TEAE) | 9 | 12
  Number of patients with Treatment Emergent Adverse Serious Event (TESAE) | 4 | 2
  Number of patients with Grade 3 or 4 Treatment Emergent Adverse Event (TEAE) | 5 | 4
  Number of patients with Treatment Emergent Adverse Event related to any of the study treatments | 8 | 11
  Number of patients with fatal events | 0 | 0
  Number of patients discontinuing for Adverse Events | 0 | 1

2. Secondary Outcome: Objective Response Rates by RECIST 1.1 and irRECIST.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Part 1: Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will then receive pembrolizumab i.v., 2mg/kg or 200mg flat dose, on day 22 (Week 3) and every 3 weeks thereafter until the end of treatment visit on day 169 (Week 24).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
- Part 2: Part 2: Patients will receive 4 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, 8 and 15) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. ONCOS-102 will be given in combination with Pembrolizumab starting on Day 22/Week 3 and every three weeks thereafter until Day 169/Week 24 or until unacceptable toxicity or clinically relevant disease progression, whichever occurs first. Pembrolizumab will be given according to institutional practice (2mg/kg or 200mg flat dose).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
Arm/Group | Part 1 | Part 2
Number analyzed (Participants) | 8 | 12
Participants
  Number of patient with Complete Response or Partial Response | 3 | 4
  Number of patients with Stable Disease or Progressive Disease | 5 | 8

3. Secondary Outcome: Changes in Immune Cell Subsets in Tumor Tissue Before and After ONCOS-102 and Pembrolizumab.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Immune Cell Subsets in Peripheral Blood Before and After ONCOS-102 and Pembrolizumab.
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Correlation of Tumour Infiltrating Lymphocytes (TILs) and Overall Response Rate (ORR).
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Progression Free Survival (PFS) Assessed by RECIST 1.1 and irRECIST.
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Benefit Rate, Defined as Any Confirmed Objective Response by RECIST 1.1 or Stable Disease.
Time Frame: 6 months
Reporting Status: Not Posted

8. Secondary Outcome: Clinical Benefit Rate, Defined as Any Objective Response by irRECIST Criteria or Immune-related Stable Disease.
Time Frame: 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in Size in Individual Lesions.
Time Frame: 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Somatic Mutational Rate and Neoepitope Burden in Tumors and Explore Relationship to Response.
Time Frame: 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in T Cell Receptor Clonality in Infiltrating and Circulating T Cells.
Time Frame: 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Gene Expression Changes in the Tumor Microenvironment and Peripheral Blood.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 27 weeks
Description: Adverse events were reported according to NCI CTCAE vs 5.0
Groups:
- Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1: Part 1: Patients will receive 3 doses of intratumoral (i.t.) injection of ONCOS-102 (days 1, 4, and 8) at 3x10^11 viral particles (VP), preceded by intravenous (i.v.) cyclophosphamide priming 1-3 days prior to day 1. They will then receive pembrolizumab i.v., 2mg/kg or 200mg flat dose, on day 22 (Week 3) and every 3 weeks thereafter until the end of treatment visit on day 169 (Week 24).
  ONCOS-102: Engineered oncolytic adenovirus expressing Granulocyte-macrophage colony stimulating factor (GM-CSF)
  Cyclophosphamide: Pre-treatment
  Pembrolizumab: PD1 blockade
Arm/Group | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1 | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/9 | 2/12
Other Adverse Events (participants affected / at risk) | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1 (N=9) | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2 (N=12)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (4)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 1 (N=9) | Experimental: ONCOS-102+Cyclophosphamide+Pembrolizumab Part 2 (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (9)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Chills (General disorders) | 5 (8) | 4 (15)
Fatigue (General disorders) | 3 (3) | 3 (3)
Injection site pain (General disorders) | 1 (2) | 3 (4)
Injection site reaction (General disorders) | 0 (0) | 3 (3)
Malaise (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 1 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (7) | 7 (23)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (8) | 3 (6)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4)
Weight decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (6) | 0 (0)
Pollakisuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 5 (7) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03003676/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT03003676/SAP_001.pdf